CLINICAL TRIAL: NCT05702307
Title: Determining the Effects of Sunflower Pasta on Glycemic Responses in Healthy Humans
Brief Title: Determining the Glycemic Effects of Sunflower Pasta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Institute of Technology and Agricultural Products (Unknown)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HRBD 60 23/06/2022
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; pasta; glycemic index; glycemic load
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: double blind (participant and outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Glucose as reference food (Experimental): Sixteen healthy, normal body weight adults after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from tagliatelle control, 5% sunflower tagliatelle, 16% sunflower tagliatelle, 16% sunflower penne, and 16% sunflower fusilli, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food
- Tagliatelle Control (Experimental): Sixteen healthy, normal body weight adults after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from tagliatelle control, 5% sunflower tagliatelle, 16% sunflower tagliatelle, 16% sunflower penne, and 16% sunflower fusilli, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Tagliatella control
- 5% sunflower tagliatelle (Experimental): Sixteen healthy, normal body weight adults after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from tagliatelle control, 5% sunflower tagliatelle, 16% sunflower tagliatelle, 16% sunflower penne, and 16% sunflower fusilli, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: 5% sunflower tagliatella
- 16% sunflower tagliatelle (Experimental): Sixteen healthy, normal body weight adults after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from tagliatelle control, 5% sunflower tagliatelle, 16% sunflower tagliatelle, 16% sunflower penne, and 16% sunflower fusilli, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: 16% sunflower tagliatella
- 16% sunflower penne (Experimental): Sixteen healthy, normal body weight adults after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from tagliatelle control, 5% sunflower tagliatelle, 16% sunflower tagliatelle, 16% sunflower penne, and 16% sunflower fusilli, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: 16% sunflower penne
- 16% sunflower fusilli (Experimental): Sixteen healthy, normal body weight adults after 12hr fast, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from tagliatelle control, 5% sunflower tagliatelle, 16% sunflower tagliatelle, 16% sunflower penne, and 16% sunflower fusilli, tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120min after food consumption. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: 16% sunflower fusilli

INTERVENTIONS:
Other: Glucose as reference food — Fifteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g glucose diluted in 300ml water, tested three times, in different visits, within 5-10min. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Glucose as reference food
Other: Tagliatella control — Fifteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from tagliatella control, tested once, in different visits, within 10min. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Tagliatelle Control
Other: 5% sunflower tagliatella — Fifteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from 5% sunflower tagliatella, tested once, in different visits, within 10min. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: 5% sunflower tagliatelle
Other: 16% sunflower tagliatella — Fifteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from 16% sunflower tagliatella, tested once, in different visits, within 10min. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: 16% sunflower tagliatelle
Other: 16% sunflower penne — Fifteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from 16% sunflower penne, tested once, in different visits, within 10min. Fingertip capillary blood glucose samples and samples from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: 16% sunflower penne
Other: 16% sunflower fusilli — Fifteen healthy, normal weight subjects after 10-14 hours fast, consumed 50g available carbohydrates from 16% sunflower fusilli, tested once, in different visits, within 10min. Fingertip capillary blood glucose samples and measurements from continuous glucose monitoring system were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: 16% sunflower fusilli

SUMMARY:
This study investigated the effects of five types of pasta on the glycemic responses

DETAILED DESCRIPTION:
This study aimed to 1.determine the glycemic index and glycemic load of five types of pasta (tagliatella control, 5% sunflower tagliatella, 16% sunflower tagliatella, 16% sunflower penne and 16% sunflower fusilli) and 2. investigate the effects of these pasta types on postprandial glycemic responses in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic men and women
* body mass index between 18 and 25 kg/m2

Exclusion Criteria:

* severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol abuse
* drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2hr
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g. hunger, satiety, desire to eat etc
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of the pasta products

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No